CLINICAL TRIAL: NCT01040403
Title: A Randomised, Double-blind, 8 Treatments, 4 Periods, Incomplete Crossover Study to Determine the Optimal Free Dose Combination of BI 1744 CL and Tiotropium Bromide (Both Delivered by the Respimat® Inhaler) After 4 Weeks Once Daily Treatment in Patients With COPD
Brief Title: Determining Optimal Free Dose Combination of Tiotropium Bromide and BI 1744 CL in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.18; 2009-014880-38 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-12-28; First posted 2009-12-29 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol

ARMS (8):
- olodaterol (BI 1744) low and placebo (Experimental): low dose inhaled olodaterol orally once daily from the Respimat inhaler
  Interventions: Drug: olodaterol (BI 1744) low; Drug: Placebo; Device: Respimat
- olodaterol (BI 1744) low and low tio (Experimental): low dose inhaled olodaterol and low dose inhaled tiotropium, both from the Respimat inhaler and once daily
  Interventions: Drug: olodaterol (BI 1744) low; Drug: low tiotropium bromide; Device: Respimat
- olodaterol (BI 1744) low and medium tio (Experimental): low dose inhaled olodaterol and medium dose inhaled tiotropium, both from the Respimat inhaler and once daily
  Interventions: Drug: olodaterol (BI 1744) low; Drug: medium tiotropium bromide; Device: Respimat
- olodaterol (BI 1744) low and high tio (Experimental): low dose inhaled olodaterol and high dose inhaled tiotropium, both from the Respimat inhaler and once daily
  Interventions: Drug: olodaterol (BI 1744) low; Drug: high tiotropium bromide; Device: Respimat
- olodaterol (BI 1744) high and placebo (Experimental): high dose inhaled olodaterol orally once daily from the Respimat inhaler
  Interventions: Drug: olodaterol (BI 1744) high; Drug: Placebo; Device: Respimat
- Olodaterol (BI 1744) high and low tio (Experimental): high dose inhaled olodaterol and low dose inhaled tiotropium, both from the Respimat inhaler and once daily
  Interventions: Drug: low tiotropium bromide; Drug: olodaterol (BI 1744) high; Device: Respimat
- Olodaterol (BI 1744) high and medium tio (Experimental): high dose inhaled olodaterol and medium dose inhaled tiotropium, both from the Respimat inhaler and once daily
  Interventions: Drug: olodaterol (BI 1744) high; Drug: medium tiotropium bromide; Device: Respimat
- Olodaterol (BI 1744) high and high tio (Experimental): high dose inhaled olodaterol and high dose inhaled tiotropium, both from the Respimat inhaler and once daily
  Interventions: Drug: olodaterol (BI 1744) high; Drug: high tiotropium bromide; Device: Respimat

INTERVENTIONS:
Drug: olodaterol (BI 1744) low — olodaterol (BI 1744) low
  Arms: olodaterol (BI 1744) low and high tio; olodaterol (BI 1744) low and low tio; olodaterol (BI 1744) low and medium tio; olodaterol (BI 1744) low and placebo
Drug: low tiotropium bromide — low tiotropium bromide
  Arms: Olodaterol (BI 1744) high and low tio; olodaterol (BI 1744) low and low tio
Drug: olodaterol (BI 1744) high — olodaterol (BI 1744) high
  Arms: Olodaterol (BI 1744) high and high tio; Olodaterol (BI 1744) high and low tio; Olodaterol (BI 1744) high and medium tio; olodaterol (BI 1744) high and placebo
Drug: medium tiotropium bromide — medium tiotropium bromide
  Arms: Olodaterol (BI 1744) high and medium tio; olodaterol (BI 1744) low and medium tio
Drug: high tiotropium bromide — high tiotropium bromide
  Arms: Olodaterol (BI 1744) high and high tio; olodaterol (BI 1744) low and high tio
Drug: Placebo — Placebo
  Arms: olodaterol (BI 1744) high and placebo; olodaterol (BI 1744) low and placebo
Device: Respimat — Respimat inhaler

SUMMARY:
The primary objective of this study is to determine the optimum once daily dose of BI 1744 CL and tiotropium in free dose combination (delivered by the Respimat inhaler) after four week treatment in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent
2. All patients must have a diagnosis of chronic obstructive pulmonary disease (COPD) must meet the following spirometric criteria:

a post-bronchodilator forced expiratory flow in 1 second (FEV1) =<30% of predicted normal and <80% of predicted normal and a post bronchodilator FEV1 / forced vital capacity (FVC) <70% at Visit 1 4. Male or female patients, 40 years of age or older. 5. Patients must be current or ex-smokers with a smoking history of more than 10 pack years

Exclusion criteria:

* Patients with a significant disease other than COPD;
* Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis;
* Patients with a history of asthma or a total blood eosinophil count >=600/mm3.
* Patients with any of the following conditions:

a diagnosis of thyrotoxicosis (due to the known class side effect profile of ß2-agonists) a diagnosis of paroxysmal tachycardia - Patients with any of the following conditions: a history of myocardial infarction within 1 year of screening visit a diagnosis of clinically relevant cardiac arrhythmia a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years

* Patients who have undergone thoracotomy with pulmonary resection
* Patients being treated with the following concomitant medications:

medications that prolong the QT/QTc interval oral Beta-adrenergics oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day

- Pregnant or nursing women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (33):
- Canada (9):
  - 1237.18.02004 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1237.18.02005 Boehringer Ingelheim Investigational Site, Grimsby, Ontario
  - 1237.18.02001 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1237.18.02008 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.18.02002 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1237.18.02003 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
  - 1237.18.02009 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 1237.18.02007 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1237.18.02011 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Germany (12):
  - 1237.18.49009 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1237.18.49012 Boehringer Ingelheim Investigational Site, Bamberg
  - 1237.18.49005 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.18.49004 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.18.49011 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.18.49010 Boehringer Ingelheim Investigational Site, Koblenz
  - 1237.18.49007 Boehringer Ingelheim Investigational Site, Mannheim
  - 1237.18.49001 Boehringer Ingelheim Investigational Site, Potsdam
  - 1237.18.49006 Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - 1237.18.49002 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1237.18.49003 Boehringer Ingelheim Investigational Site, Weinheim
  - 1237.18.49008 Boehringer Ingelheim Investigational Site, Wiesloch
- Netherlands (8):
  - 1237.18.31004 Boehringer Ingelheim Investigational Site, Almelo
  - 1237.18.31006 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1237.18.31008 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1237.18.31001 Boehringer Ingelheim Investigational Site, Groningen
  - 1237.18.31007 Boehringer Ingelheim Investigational Site, Hengelo
  - 1237.18.31005 Boehringer Ingelheim Investigational Site, Hoorn
  - 1237.18.31002 Boehringer Ingelheim Investigational Site, Veldhoven
  - 1237.18.31003 Boehringer Ingelheim Investigational Site, Zutphen
- Sweden (4):
  - 1237.18.46003 Boehringer Ingelheim Investigational Site, Boden
  - 1237.18.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1237.18.46001 Boehringer Ingelheim Investigational Site, Lund
  - 1237.18.46004 Boehringer Ingelheim Investigational Site, Stockholm

REFERENCES:
- [Derived] Aalbers R, Maleki-Yazdi MR, Hamilton A, Waitere-Wijker S, Zhao Y, Amatto VC, Schmidt O, Bjermer L. Randomized, Double-Blind, Dose-Finding Study for Tiotropium when Added to Olodaterol, Administered via the Respimat(R) Inhaler in Patients with Chronic Obstructive Pulmonary Disease. Adv Ther. 2015 Sep;32(9):809-22. doi: 10.1007/s12325-015-0239-8. Epub 2015 Sep 24. PMID 26404912

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, 4-period incomplete cross-over trial. 233 patients were randomized to one of 14 treatment sequences and 232 of them were treated. It was a double-blind trial in which each treatment period lasted 4 weeks with a washout period of 21 days between each.
Groups:
- Overall Study: A randomised, double-blind, 8 treatment, 4 period, incomplete crossover study. Each treatment period was separated by a washout period of 3 weeks. The 8 treatments, administered by oral inhalation from separate Respimat inhalers, once daily, in the morning, were:
  * Olodaterol 5 µg and placebo
  * Tiotropium 1.25 µg and Olodaterol 5 µg free combination inhalation solution
  * Tiotropium 2.5 µg and Olodaterol 5 µg free combination inhalation solution
  * Tiotropium 5 µg and Olodaterol 5 µg free combination inhalation solution
  * Olodaterol 10 µg and placebo
  * Tiotropium 1.25 µg and Olodaterol 10 µg free combination inhalation solution
  * Tiotropium 2.5 µg and Olodaterol 10 µg free combination inhalation solution
  * Tiotropium 5 µg and Olodaterol 10 µg free combination inhalation solution
Period: Overall Study
Arm/Group | Overall Study
Started | 233
Completed Olo 5 | 106
Completed T+O 1.25/5 | 105
Completed T+O 2.5/5 | 111
Completed T+O 5/5 | 106
Completed Olo 10 | 109
Completed T+O 1.25/10 | 106
Completed T+O 2.5/10 | 110
Completed T+O 5/10 | 107
Completed | 213 (All treatment periods)
Not Completed | 20
Not completed — Adverse Event | 10
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 1
Not completed — Not treated | 1
Not completed — Other reason not defined above | 6

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) which comprised all patients who were dispensed study medication and were documented to have taken at least 1 dose of investigational treatment.
Arm/Group | Overall Study
Number analyzed (Participants) | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 133

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 Response
Description: Adjusted means of the trough forced expiratory volume in one second (FEV1) response (L) after four weeks treatment. The trough was defined as the mean of the 1 h pre-dose and 10 min pre-dose measurements on day 29. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 hour pre-dose and 10 minutes pre-dose on day 29
Population: Full Analysis Set (FAS) which comprised all patients in the treated set who provided baseline (study baseline) data and at least 1 on-treatment efficacy value for the primary endpoint after 4 weeks on treatment.
Measure: Mean (Standard Deviation); unit: Litres
Groups:
- Olo 5: Oral inhalation of Olodaterol 5 µg and placebo (Olodaterol: 2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- T+O 1.25/5: Oral inhalation of Tiotropium 1.25 µg and Olodaterol 5 µg (Tiotropium: 0.625 µg per actuation and Olodaterol: 2.5 µg per actuation) as free combination inhalation solution, 2 puffs from separate Respimat inhalers, once daily, in the morning.
- T+O 2.5/5: Oral inhalation of Tiotropium 2.5 µg and Olodaterol 5 µg (Tiotropium: 1.25 µg per actuation and Olodaterol: 2.5 µg per actuation), as free combination inhalation solution, 2 puffs from separate Respimat inhalers, once daily, in the morning.
- T+O 5/5: Oral inhalation of Tiotropium 5 µg and Olodaterol 5 µg (Tiotropium and Olodaterol: 2.5 µg per actuation), as free combination inhalation solution, 2 puffs from separate Respimat inhalers, once daily, in the morning.
- Olo 10: Oral inhalation of Olodaterol 10 µg and placebo (Olodaterol: 5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- T+O 1.25/10: Oral inhalation of Tiotropium 1.25 µg and Olodaterol 10 µg (Tiotropium: 0.625 µg per actuation and Olodaterol: 5 µg per actuation), as free combination inhalation solution, 2 puffs from separate Respimat inhalers, once daily, in the morning.
- T+O 2.5/10: Oral inhalation of Tiotropium 2.5 µg and Olodaterol 10 µg (Tiotropium: 1.25 µg per actuation and Olodaterol: 5 µg per actuation), as free combination inhalation solution, 2 puffs from separate Respimat inhalers, once daily, in the morning
- T+O 5/10: Oral inhalation of Tiotropium 5 µg and Olodaterol 10 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 5 µg per actuation), as free combination inhalation solution, 2 puffs from separate Respimat inhalers, once daily, in the morning.
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.071 (0.018) | 0.125 (0.018) | 0.136 (0.018) | 0.155 (0.018) | 0.083 (0.018) | 0.134 (0.018) | 0.166 (0.018) | 0.163 (0.018)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.054, 95% CI 2-sided [0.016 to 0.092], Standard Error of Mean 0.019 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.065, 95% CI 2-sided [0.027 to 0.103], Standard Error of Mean 0.019 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.084, 95% CI 2-sided [0.046 to 0.122], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.027 to 0.049], Standard Error of Mean 0.019 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.008 to 0.069], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.019, 95% CI 2-sided [-0.019 to 0.058], Standard Error of Mean 0.019 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.051, 95% CI 2-sided [0.013 to 0.089], Standard Error of Mean 0.019 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.083, 95% CI 2-sided [0.045 to 0.122], Standard Error of Mean 0.019 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.080, 95% CI 2-sided [0.042 to 0.119], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.033, 95% CI 2-sided [-0.006 to 0.071], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.009 to 0.068], Standard Error of Mean 0.019 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.041 to 0.035], Standard Error of Mean 0.019 — Difference calculated as T+O 5/10 minus T+O 2.5/10

2. Secondary Outcome: Trough Forced Vital Capacity (FVC) Response
Description: Adjusted means of trough FVC (forced vital capacity) response [L] after 4 weeks treatment. The trough was defined as the mean of the 1 h pre-dose and 10 min pre-dose measurements on day 29. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 hour pre-dose and 10 minutes pre-dose on day 29
Population: FAS which included all patients who were dispensed study medication and who provided baseline and at least 1 on-treatment efficacy value for the primary endpoint after 4 weeks on treatment.
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.114 (0.029) | 0.214 (0.029) | 0.234 (0.029) | 0.215 (0.029) | 0.122 (0.029) | 0.253 (0.029) | 0.253 (0.029) | 0.249 (0.029)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.099, 95% CI 2-sided [0.040 to 0.159], Standard Error of Mean 0.030 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.120, 95% CI 2-sided [0.061 to 0.179], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.100, 95% CI 2-sided [0.041 to 0.160], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.039 to 0.079], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.059 to 0.061], Standard Error of Mean 0.031 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.019, 95% CI 2-sided [-0.079 to 0.040], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.071 to 0.190], Standard Error of Mean 0.030 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.072 to 0.191], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.127, 95% CI 2-sided [0.067 to 0.187], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.059 to 0.061], Standard Error of Mean 0.031 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.063 to 0.056], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.064 to 0.055], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus T+O 2.5/10

3. Secondary Outcome: FEV1 AUC 0-3h and FEV1 AUC 0-6h Response
Description: Adjusted means of forced expiratory volume in one second (FEV1) area under the curve (AUC) 0-3 hour and AUC 0-6 hour responses [L] after 4 weeks treatment calculated using the trapezoidal rule, divided by the duration (3 h, 6 h) to report in litres. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post dose for AUC0-3h and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h 4 h, 5 h, 6 h postdose for AUC0-6h on day 29
Population: FAS
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres
  AUC 0-3h | 0.183 (0.020) | 0.258 (0.020) | 0.280 (0.020) | 0.302 (0.020) | 0.191 (0.020) | 0.288 (0.020) | 0.319 (0.020) | 0.334 (0.020)
  AUC 0-6h | 0.188 (0.020) | 0.267 (0.020) | 0.287 (0.020) | 0.307 (0.020) | 0.198 (0.020) | 0.296 (0.020) | 0.320 (0.020) | 0.342 (0.020)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.075, 95% CI 2-sided [0.035 to 0.114], Standard Error of Mean 0.020 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.097, 95% CI 2-sided [0.057 to 0.137], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.119, 95% CI 2-sided [0.079 to 0.159], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.017 to 0.062], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [0.004 to 0.085], Standard Error of Mean 0.021 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.018 to 0.062], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.097, 95% CI 2-sided [0.057 to 0.137], Standard Error of Mean 0.020 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.128, 95% CI 2-sided [0.088 to 0.168], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.143, 95% CI 2-sided [0.103 to 0.183], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.009 to 0.071], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [0.006 to 0.086], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.015, 95% CI 2-sided [-0.025 to 0.055], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus T+O 2.5/10
Statistical Analysis 13: Comparison: Olo 5 vs T+O 1.25/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [0.040 to 0.117], Standard Error of Mean 0.020 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 14: Comparison: Olo 5 vs T+O 2.5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.099, 95% CI 2-sided [0.060 to 0.137], Standard Error of Mean 0.019 — difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 15: Comparison: Olo 5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [0.080 to 0.157], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 16: Comparison: T+O 1.25/5 vs T+O 2.5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.018 to 0.058], Standard Error of Mean 0.019 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 17: Comparison: T+O 1.25/5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [0.001 to 0.079], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 18: Comparison: T+O 2.5/5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.020, 95% CI 2-sided [-0.019 to 0.058], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 19: Comparison: Olo 10 vs T+O 1.25/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [0.060 to 0.136], Standard Error of Mean 0.020 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 20: Comparison: Olo 10 vs T+O 2.5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [0.083 to 0.159], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 21: Comparison: Olo 10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [0.105 to 0.182], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 22: Comparison: T+O 1.25/10 vs T+O 2.5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.016 to 0.062], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 23: Comparison: T+O 1.25/10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [0.007 to 0.084], Standard Error of Mean 0.019 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 24: Comparison: T+O 2.5/10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [-0.016 to 0.061], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus T+O 2.5/10

4. Secondary Outcome: FEV1 AUC 0-3h Response After the First Dose
Description: Adjusted means of Forced Expiratory Volume in One Second (FEV1) Area Under Curve (AUC) 0-3h response [L] after the first dose, calculated using the trapezoidal rule, divided by the duration (3 hours) to report in litres. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 1
Population: FAS
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.204 (0.017) | 0.181 (0.017) | 0.209 (0.017) | 0.205 (0.017) | 0.188 (0.017) | 0.227 (0.017) | 0.219 (0.017) | 0.230 (0.017)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.023, 95% CI 2-sided [-0.058 to 0.012], Standard Error of Mean 0.018 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.005, 95% CI 2-sided [-0.029 to 0.040], Standard Error of Mean 0.018 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.001, 95% CI 2-sided [-0.034 to 0.036], Standard Error of Mean 0.018 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.006 to 0.063], Standard Error of Mean 0.018 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.011 to 0.059], Standard Error of Mean 0.018 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.039 to 0.031], Standard Error of Mean 0.018 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.039, 95% CI 2-sided [0.004 to 0.073], Standard Error of Mean 0.018 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.004 to 0.066], Standard Error of Mean 0.018 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.041, 95% CI 2-sided [0.006 to 0.076], Standard Error of Mean 0.018 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.043 to 0.027], Standard Error of Mean 0.018 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.032 to 0.037], Standard Error of Mean 0.018 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.010, 95% CI 2-sided [-0.025 to 0.045], Standard Error of Mean 0.018 — Difference calculated as T+O 5/10 minus T+O 2.5/10

5. Secondary Outcome: FEV1 Peak 0-3h Response
Description: Adjusted means of the FEV1 peak value over the time from 0 to 3 hours (peak 0-3h) response [L] after 4 weeks of treatment. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.264 (0.023) | 0.353 (0.023) | 0.355 (0.023) | 0.379 (0.023) | 0.267 (0.023) | 0.374 (0.023) | 0.399 (0.023) | 0.412 (0.023)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.089, 95% CI 2-sided [0.041 to 0.138], Standard Error of Mean 0.025 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.091, 95% CI 2-sided [0.043 to 0.139], Standard Error of Mean 0.024 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.115, 95% CI 2-sided [0.066 to 0.164], Standard Error of Mean 0.025 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.046 to 0.050], Standard Error of Mean 0.025 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.026, 95% CI 2-sided [-0.023 to 0.074], Standard Error of Mean 0.025 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.025 to 0.072], Standard Error of Mean 0.025 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.107, 95% CI 2-sided [0.059 to 0.156], Standard Error of Mean 0.025 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.132, 95% CI 2-sided [0.084 to 0.181], Standard Error of Mean 0.025 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.145, 95% CI 2-sided [0.096 to 0.193], Standard Error of Mean 0.025 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.025, 95% CI 2-sided [-0.024 to 0.074], Standard Error of Mean 0.025 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.038, 95% CI 2-sided [-0.010 to 0.086], Standard Error of Mean 0.025 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.036 to 0.061], Standard Error of Mean 0.025 — Difference calculated as T+O 5/10 minus T+O 2.5/10

6. Secondary Outcome: FEV1 Peak 0-3h Response After the First Dose
Description: Adjusted means of the FEV1 peak 0-3h response [L] after the first dose of treatment. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 1
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.287 (0.019) | 0.267 (0.019) | 0.300 (0.019) | 0.298 (0.019) | 0.270 (0.019) | 0.324 (0.019) | 0.315 (0.019) | 0.317 (0.019)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.019, 95% CI 2-sided [-0.059 to 0.020], Standard Error of Mean 0.020 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.026 to 0.053], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.012, 95% CI 2-sided [-0.028 to 0.051], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.033, 95% CI 2-sided [-0.006 to 0.072], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.031, 95% CI 2-sided [-0.009 to 0.071], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.002, 95% CI 2-sided [-0.041 to 0.037], Standard Error of Mean 0.020 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.054, 95% CI 2-sided [0.015 to 0.093], Standard Error of Mean 0.020 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.045, 95% CI 2-sided [0.006 to 0.084], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.047, 95% CI 2-sided [0.008 to 0.087], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.009, 95% CI 2-sided [-0.049 to 0.031], Standard Error of Mean 0.020 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.046 to 0.033], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.037 to 0.042], Standard Error of Mean 0.020 — Difference calculated as T+O 5/10 minus T+O 2.5/10

7. Secondary Outcome: FVC AUC 0-3h and FEV1 AUC 0-6h Responses
Description: Adjusted means of the FVC AUC 0-3h and AUC 0-6h responses [L] after 4 weeks of treatment, calculated using the trapezoidal rule, divided by the duration (3 h, 6 h) to report in litres. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: as for outcome 3
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres
  AUC 0-3h | 0.278 (0.032) | 0.422 (0.032) | 0.429 (0.032) | 0.410 (0.032) | 0.279 (0.032) | 0.455 (0.032) | 0.454 (0.032) | 0.479 (0.032)
  AUC 0-6h | 0.282 (0.032) | 0.421 (0.032) | 0.432 (0.032) | 0.414 (0.032) | 0.277 (0.032) | 0.466 (0.032) | 0.456 (0.032) | 0.490 (0.032)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.143, 95% CI 2-sided [0.084 to 0.202], Standard Error of Mean 0.030 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.151, 95% CI 2-sided [0.092 to 0.210], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.072 to 0.191], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.051 to 0.066], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.071 to 0.048], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.020, 95% CI 2-sided [-0.079 to 0.039], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.175, 95% CI 2-sided [0.116 to 0.234], Standard Error of Mean 0.030 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.175, 95% CI 2-sided [0.116 to 0.234], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.200, 95% CI 2-sided [0.140 to 0.259], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.000, 95% CI 2-sided [-0.060 to 0.059], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.035 to 0.083], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.035 to 0.083], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus T+O 2.5/10
Statistical Analysis 13: Comparison: Olo 5 vs T+O 1.25/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.139, 95% CI 2-sided [0.081 to 0.197], Standard Error of Mean 0.029 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 14: Comparison: Olo 5 vs T+O 2.5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.150, 95% CI 2-sided [0.092 to 0.207], Standard Error of Mean 0.029 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 15: Comparison: Olo 5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.073 to 0.189], Standard Error of Mean 0.029 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 16: Comparison: T+O 1.25/5 vs T+O 2.5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.011, 95% CI 2-sided [-0.047 to 0.068], Standard Error of Mean 0.029 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 17: Comparison: T+O 1.25/5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.066 to 0.051], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 18: Comparison: T+O 2.5/5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.018, 95% CI 2-sided [-0.076 to 0.039], Standard Error of Mean 0.029 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 19: Comparison: Olo 10 vs T+O 1.25/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.189, 95% CI 2-sided [0.131 to 0.247], Standard Error of Mean 0.029 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 20: Comparison: Olo 10 vs T+O 2.5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.179, 95% CI 2-sided [0.121 to 0.236], Standard Error of Mean 0.029 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 21: Comparison: Olo 10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.213, 95% CI 2-sided [0.155 to 0.271], Standard Error of Mean 0.029 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 22: Comparison: T+O 1.25/10 vs T+O 2.5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.010, 95% CI 2-sided [-0.069 to 0.048], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 23: Comparison: T+O 1.25/10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.033 to 0.082], Standard Error of Mean 0.029 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 24: Comparison: T+O 2.5/10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.035, 95% CI 2-sided [-0.023 to 0.092], Standard Error of Mean 0.029 — Difference calculated as T+O 5/10 minus T+O 2.5/10

8. Secondary Outcome: FVC AUC 0-3h Response After First Dose
Description: Adjusted means of the FVC AUC 0-3h response [L] after first dose, calculated using the trapezoidal rule, divided by the duration (3 hours) to report in litres. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on days 1
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.333 (0.029) | 0.285 (0.029) | 0.326 (0.029) | 0.319 (0.030) | 0.303 (0.029) | 0.393 (0.030) | 0.363 (0.029) | 0.359 (0.029)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.048, 95% CI 2-sided [-0.106 to 0.010], Standard Error of Mean 0.029 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.065 to 0.051], Standard Error of Mean 0.029 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.014, 95% CI 2-sided [-0.072 to 0.044], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.041, 95% CI 2-sided [-0.017 to 0.099], Standard Error of Mean 0.029 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.024 to 0.093], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.007, 95% CI 2-sided [-0.065 to 0.051], Standard Error of Mean 0.030 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.090, 95% CI 2-sided [0.032 to 0.148], Standard Error of Mean 0.030 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [0.001 to 0.118], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.056, 95% CI 2-sided [-0.002 to 0.114], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.031, 95% CI 2-sided [-0.089 to 0.028], Standard Error of Mean 0.030 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.034, 95% CI 2-sided [-0.092 to 0.024], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.062 to 0.055], Standard Error of Mean 0.030 — Difference calculated as T+O 5/10 minus T+O 2.5/10

9. Secondary Outcome: FVC Peak 0-3h Response
Description: Adjusted means of the FVC peak 0-3h response [L] after 4 weeks of treatment. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.415 (0.035) | 0.570 (0.035) | 0.563 (0.035) | 0.542 (0.035) | 0.411 (0.035) | 0.585 (0.035) | 0.593 (0.035) | 0.615 (0.035)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.155, 95% CI 2-sided [0.087 to 0.223], Standard Error of Mean 0.035 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.147, 95% CI 2-sided [0.079 to 0.215], Standard Error of Mean 0.035 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.127, 95% CI 2-sided [0.058 to 0.195], Standard Error of Mean 0.035 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.008, 95% CI 2-sided [-0.075 to 0.060], Standard Error of Mean 0.035 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.028, 95% CI 2-sided [-0.097 to 0.041], Standard Error of Mean 0.035 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.020, 95% CI 2-sided [-0.089 to 0.048], Standard Error of Mean 0.035 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.174, 95% CI 2-sided [0.106 to 0.242], Standard Error of Mean 0.035 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.182, 95% CI 2-sided [0.113 to 0.250], Standard Error of Mean 0.035 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.204, 95% CI 2-sided [0.135 to 0.272], Standard Error of Mean 0.035 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.061 to 0.076], Standard Error of Mean 0.035 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.030, 95% CI 2-sided [-0.038 to 0.098], Standard Error of Mean 0.035 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.046 to 0.090], Standard Error of Mean 0.035 — Difference calculated as T+O 5/10 minus T+O 2.5/10

10. Secondary Outcome: FVC Peak 0-3h Response After the First Dose
Description: Adjusted mean of the FVC peak 0-3h response [L] after the first dose. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 1
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres | 0.473 (0.031) | 0.423 (0.031) | 0.481 (0.031) | 0.462 (0.032) | 0.436 (0.031) | 0.547 (0.032) | 0.517 (0.031) | 0.505 (0.031)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.051, 95% CI 2-sided [-0.114 to 0.013], Standard Error of Mean 0.032 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.008, 95% CI 2-sided [-0.055 to 0.071], Standard Error of Mean 0.032 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.011, 95% CI 2-sided [-0.074 to 0.053], Standard Error of Mean 0.032 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.059, 95% CI 2-sided [-0.004 to 0.122], Standard Error of Mean 0.032 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.040, 95% CI 2-sided [-0.024 to 0.104], Standard Error of Mean 0.033 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.019, 95% CI 2-sided [-0.082 to 0.045], Standard Error of Mean 0.032 — Difference calculated as T+O 5/5 minus +O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.111, 95% CI 2-sided [0.047 to 0.174], Standard Error of Mean 0.032 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.081, 95% CI 2-sided [0.017 to 0.144], Standard Error of Mean 0.032 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.069, 95% CI 2-sided [0.005 to 0.132], Standard Error of Mean 0.032 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.030, 95% CI 2-sided [-0.094 to 0.034], Standard Error of Mean 0.033 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.042, 95% CI 2-sided [-0.105 to 0.021], Standard Error of Mean 0.032 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.012, 95% CI 2-sided [-0.075 to 0.052], Standard Error of Mean 0.032 — Difference calculated as T+O 5/10 minus T+O 2.5/10

11. Secondary Outcome: PEF AUC 0-3h and AUC 0-6h Responses
Description: Adjusted means of the Peak Expiratory Flow (PEF) AUC 0-3h and AUC 0-6h responses in Litres / minute (L/min) after 4 weeks of treatment, calculated using the trapezoidal rule, divided by the duration (3 h, 6 h) to report in litres. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: as for outcome 3
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
L/min
  AUC 0-3h | 25.542 (4.190) | 44.301 (4.202) | 50.698 (4.167) | 55.346 (4.234) | 29.713 (4.183) | 48.032 (4.218) | 53.224 (4.192) | 52.531 (4.205)
  AUC 0-6h | 28.071 (4.125) | 46.822 (4.136) | 54.081 (4.104) | 57.418 (4.166) | 31.831 (4.119) | 51.485 (4.151) | 54.593 (4.127) | 57.367 (4.139)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 18.759, 95% CI 2-sided [10.533 to 26.985], Standard Error of Mean 4.189 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 25.157, 95% CI 2-sided [16.962 to 33.351], Standard Error of Mean 4.173 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 29.804, 95% CI 2-sided [21.526 to 38.082], Standard Error of Mean 4.216 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 6.398, 95% CI 2-sided [-1.796 to 14.592], Standard Error of Mean 4.173 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 11.046, 95% CI 2-sided [2.721 to 19.370], Standard Error of Mean 4.239 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.648, 95% CI 2-sided [-3.608 to 12.903], Standard Error of Mean 4.204 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 18.318, 95% CI 2-sided [10.068 to 26.568], Standard Error of Mean 4.201 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 23.511, 95% CI 2-sided [15.270 to 31.752], Standard Error of Mean 4.197 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 22.817, 95% CI 2-sided [14.543 to 31.092], Standard Error of Mean 4.214 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.193, 95% CI 2-sided [-3.115 to 13.500], Standard Error of Mean 4.230 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.499, 95% CI 2-sided [-3.719 to 12.717], Standard Error of Mean 4.185 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; AUC 0-3h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.694, 95% CI 2-sided [-8.941 to 7.554], Standard Error of Mean 4.200 — Difference calculated as T+O 5/10 minus T+O 2.5/10
Statistical Analysis 13: Comparison: Olo 5 vs T+O 1.25/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 18.751, 95% CI 2-sided [10.870 to 26.632], Standard Error of Mean 4.013 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 14: Comparison: Olo 5 vs T+O 2.5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 26.009, 95% CI 2-sided [18.158 to 33.860], Standard Error of Mean 3.998 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 15: Comparison: Olo 5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 29.347, 95% CI 2-sided [21.416 to 37.278], Standard Error of Mean 4.039 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 16: Comparison: T+O 1.25/5 vs T+O 2.5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 7.259, 95% CI 2-sided [-0.592 to 15.109], Standard Error of Mean 3.998 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 17: Comparison: T+O 1.25/5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 10.596, 95% CI 2-sided [2.621 to 18.571], Standard Error of Mean 4.061 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 18: Comparison: T+O 2.5/5 vs T+O 5/5; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.337, 95% CI 2-sided [-4.572 to 11.247], Standard Error of Mean 4.028 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 19: Comparison: Olo 10 vs T+O 1.25/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 19.654, 95% CI 2-sided [11.750 to 27.558], Standard Error of Mean 4.025 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 20: Comparison: Olo 10 vs T+O 2.5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 22.762, 95% CI 2-sided [14.866 to 30.659], Standard Error of Mean 4.021 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 21: Comparison: Olo 10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 25.536, 95% CI 2-sided [17.607 to 33.464], Standard Error of Mean 4.038 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 22: Comparison: T+O 1.25/10 vs T+O 2.5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.108, 95% CI 2-sided [-4.852 to 11.067], Standard Error of Mean 4.053 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 23: Comparison: T+O 1.25/10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.881, 95% CI 2-sided [-1.991 to 13.754], Standard Error of Mean 4.009 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 24: Comparison: T+O 2.5/10 vs T+O 5/10; AUC 0-6h; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.773, 95% CI 2-sided [-5.129 to 10.675], Standard Error of Mean 4.024 — Difference calculated as T+O 5/10 minus T+O 2.5/10

12. Secondary Outcome: PEF AUC 0-3h Response After the First Dose
Description: Adjusted means of the Area under the curve from 0 to 3 h response in Litres / minutes of the peak expiratory flow after the first dose, calculated using the trapezoidal rule, divided by the duration (3 hours) to report in litres. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 1
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
L/min | 30.575 (4.047) | 32.891 (4.050) | 35.053 (4.022) | 35.243 (4.084) | 31.724 (4.040) | 33.213 (4.079) | 34.987 (4.051) | 38.846 (4.065)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.316, 95% CI 2-sided [-6.268 to 10.900], Standard Error of Mean 4.371 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.478, 95% CI 2-sided [-4.088 to 13.044], Standard Error of Mean 4.362 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.668, 95% CI 2-sided [-3.978 to 13.314], Standard Error of Mean 4.403 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.162, 95% CI 2-sided [-6.379 to 10.702], Standard Error of Mean 4.349 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.352, 95% CI 2-sided [-6.326 to 11.029], Standard Error of Mean 4.419 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.190, 95% CI 2-sided [-8.430 to 8.810], Standard Error of Mean 4.390 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.488, 95% CI 2-sided [-7.136 to 10.113], Standard Error of Mean 4.392 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.262, 95% CI 2-sided [-5.350 to 11.875], Standard Error of Mean 4.386 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 7.121, 95% CI 2-sided [-1.535 to 15.778], Standard Error of Mean 4.408 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.774, 95% CI 2-sided [-6.910 to 10.458], Standard Error of Mean 4.423 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.663, 95% CI 2-sided [-2.970 to 14.236], Standard Error of Mean 4.381 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.859, 95% CI 2-sided [-4.786 to 12.504], Standard Error of Mean 4.403 — Difference calculated as T+O 5/10 minus T+O 2.5/10

13. Secondary Outcome: PEF Peak 0-3h Response
Description: Adjusted means of the peak expiratory flow from 0 to 3 hours (PEF peak 0-3h) response in L/min after 4 weeks of treatment. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 29
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
L/min | 46.010 (4.566) | 64.693 (4.581) | 69.610 (4.538) | 76.108 (4.620) | 49.025 (4.557) | 66.767 (4.600) | 73.140 (4.569) | 74.120 (4.584)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 18.682, 95% CI 2-sided [9.161 to 28.204], Standard Error of Mean 4.849 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 23.599, 95% CI 2-sided [14.116 to 33.083], Standard Error of Mean 4.830 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 30.097, 95% CI 2-sided [20.517 to 39.677], Standard Error of Mean 4.879 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.917, 95% CI 2-sided [-4.568 to 14.402], Standard Error of Mean 4.830 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 11.415, 95% CI 2-sided [1.780 to 21.050], Standard Error of Mean 4.907 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 6.498, 95% CI 2-sided [-3.057 to 16.053], Standard Error of Mean 4.866 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 17.742, 95% CI 2-sided [8.194 to 27.290], Standard Error of Mean 4.862 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 24.115, 95% CI 2-sided [14.580 to 33.651], Standard Error of Mean 4.856 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 25.095, 95% CI 2-sided [15.520 to 34.670], Standard Error of Mean 4.876 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 6.373, 95% CI 2-sided [-3.240 to 15.986], Standard Error of Mean 4.896 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 7.353, 95% CI 2-sided [-2.161 to 16.866], Standard Error of Mean 4.845 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.980, 95% CI 2-sided [-8.566 to 10.525], Standard Error of Mean 4.861 — Difference calculated as T+O 5/10 minus T+O 2.5/10

14. Secondary Outcome: PEF Peak 0-3h Response After the First Dose
Description: Adjusted means of the Peak Expiratory flow from 0 to 3 hours response in L/min after the first dose of treatment. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 5 min, 30 min, 1 h, 2 h, 3 h post-dose on day 1
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
L/min | 52.129 (4.363) | 53.298 (4.366) | 56.565 (4.335) | 57.318 (4.406) | 51.980 (4.355) | 54.966 (4.400) | 56.896 (4.367) | 59.412 (4.370)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.170, 95% CI 2-sided [-8.360 to 10.699], Standard Error of Mean 4.853 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.436, 95% CI 2-sided [-5.073 to 13.945], Standard Error of Mean 4.843 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.189, 95% CI 2-sided [-4.407 to 14.785], Standard Error of Mean 4.887 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 3.267, 95% CI 2-sided [-6.214 to 12.747], Standard Error of Mean 4.828 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.020, 95% CI 2-sided [-5.610 to 13.650], Standard Error of Mean 4.904 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.753, 95% CI 2-sided [-8.816 to 10.322], Standard Error of Mean 4.873 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.986, 95% CI 2-sided [-6.589 to 12.561], Standard Error of Mean 4.876 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.916, 95% CI 2-sided [-4.643 to 14.475], Standard Error of Mean 4.868 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 7.432, 95% CI 2-sided [-2.154 to 17.019], Standard Error of Mean 4.882 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 1.930, 95% CI 2-sided [-7.708 to 11.568], Standard Error of Mean 4.909 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 4.446, 95% CI 2-sided [-5.085 to 13.978], Standard Error of Mean 4.854 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.517, 95% CI 2-sided [-7.046 to 12.079], Standard Error of Mean 4.870 — Difference calculated as T+O 5/10 minus T+O 2.5/10

15. Secondary Outcome: Individual FEV1 Measurements at Each Time Point on Day 29
Description: Adjusted means of the FEV1 measurements [L] at each time point on day 29. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 0 min, 5 min, 30 min, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h post-dose on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres
  Timepoint -1:00 hr response | 1.410 (0.018) | 1.464 (0.018) | 1.481 (0.018) | 1.491 (0.018) | 1.414 (0.018) | 1.467 (0.018) | 1.504 (0.018) | 1.500 (0.018)
  Timepoint -0:10 hr response | 1.431 (0.020) | 1.487 (0.020) | 1.488 (0.020) | 1.516 (0.020) | 1.447 (0.020) | 1.498 (0.020) | 1.526 (0.020) | 1.527 (0.020)
  Timepoint 0:00 hr response | 1.419 (0.018) | 1.473 (0.018) | 1.484 (0.018) | 1.503 (0.018) | 1.431 (0.018) | 1.482 (0.018) | 1.514 (0.018) | 1.511 (0.018)
  Timepoint 0:05 hr response | 1.483 (0.022) | 1.555 (0.022) | 1.553 (0.022) | 1.563 (0.022) | 1.491 (0.022) | 1.576 (0.022) | 1.593 (0.022) | 1.601 (0.022)
  Timepoint 0:30 hr response | 1.516 (0.021) | 1.570 (0.021) | 1.597 (0.021) | 1.630 (0.021) | 1.524 (0.021) | 1.605 (0.021) | 1.643 (0.021) | 1.660 (0.021)
  Timepoint 1:00 hr response | 1.521 (0.021) | 1.595 (0.021) | 1.622 (0.021) | 1.633 (0.021) | 1.527 (0.021) | 1.627 (0.021) | 1.658 (0.021) | 1.675 (0.021)
  Timepoint 2:00 hr response | 1.552 (0.021) | 1.625 (0.021) | 1.656 (0.021) | 1.687 (0.022) | 1.556 (0.021) | 1.661 (0.021) | 1.699 (0.021) | 1.711 (0.021)
  Timepoint 3:00 hr response | 1.553 (0.022) | 1.648 (0.022) | 1.659 (0.022) | 1.671 (0.022) | 1.567 (0.022) | 1.671 (0.022) | 1.690 (0.022) | 1.716 (0.022)
  Timepoint 4:00 hr response | 1.543 (0.021) | 1.621 (0.021) | 1.654 (0.021) | 1.659 (0.021) | 1.563 (0.021) | 1.663 (0.021) | 1.676 (0.021) | 1.708 (0.021)
  Timepoint 5:00 hr response | 1.549 (0.021) | 1.622 (0.021) | 1.626 (0.021) | 1.654 (0.021) | 1.540 (0.021) | 1.640 (0.021) | 1.655 (0.021) | 1.688 (0.021)
  Timepoint 6:00 hr response | 1.517 (0.022) | 1.605 (0.022) | 1.631 (0.021) | 1.647 (0.022) | 1.547 (0.022) | 1.636 (0.022) | 1.656 (0.022) | 1.687 (0.022)

16. Secondary Outcome: Individual FVC Measurements at Each Time Point on Day 29
Description: Adjusted means of the FVC measurements [L] at each time point on day 29. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 0 min, 5 min, 30 min, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h post-dose on day 29
Population: FAS
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
Litres
  Timepoint -1:00 hr response | 2.877 (0.029) | 2.961 (0.029) | 2.996 (0.029) | 2.954 (0.029) | 2.877 (0.029) | 3.006 (0.029) | 3.012 (0.029) | 3.007 (0.029)
  Timepoint -0:10 hr response | 2.891 (0.032) | 3.007 (0.032) | 3.009 (0.031) | 3.012 (0.032) | 2.904 (0.032) | 3.036 (0.032) | 3.032 (0.032) | 3.032 (0.032)
  Timepoint 0:00 hr response | 2.882 (0.029) | 2.981 (0.029) | 3.002 (0.029) | 2.982 (0.029) | 2.889 (0.029) | 3.020 (0.029) | 3.020 (0.029) | 3.016 (0.029)
  Timepoint 0:05 hr response | 2.999 (0.033) | 3.130 (0.033) | 3.120 (0.033) | 3.087 (0.033) | 3.009 (0.033) | 3.141 (0.033) | 3.147 (0.033) | 3.148 (0.033)
  Timepoint 0:30 hr response | 3.018 (0.033) | 3.171 (0.033) | 3.145 (0.033) | 3.172 (0.034) | 3.019 (0.033) | 3.190 (0.034) | 3.192 (0.033) | 3.219 (0.033)
  Timepoint 1:00 hr response | 3.036 (0.034) | 3.174 (0.034) | 3.190 (0.034) | 3.162 (0.034) | 3.032 (0.034) | 3.204 (0.034) | 3.215 (0.034) | 3.239 (0.034)
  Timepoint 2:00 hr response | 3.077 (0.034) | 3.216 (0.034) | 3.234 (0.034) | 3.208 (0.035) | 3.071 (0.034) | 3.258 (0.035) | 3.249 (0.034) | 3.275 (0.034)
  Timepoint 3:00 hr response | 3.067 (0.035) | 3.222 (0.035) | 3.233 (0.035) | 3.200 (0.036) | 3.081 (0.035) | 3.264 (0.036) | 3.267 (0.035) | 3.303 (0.035)
  Timepoint 4:00 hr response | 3.054 (0.035) | 3.181 (0.035) | 3.204 (0.034) | 3.183 (0.035) | 3.054 (0.034) | 3.266 (0.035) | 3.227 (0.035) | 3.281 (0.035)
  Timepoint 5:00 hr response | 3.061 (0.035) | 3.193 (0.035) | 3.188 (0.035) | 3.178 (0.035) | 3.019 (0.035) | 3.222 (0.035) | 3.214 (0.035) | 3.252 (0.035)
  Timepoint 6:00 hr response | 3.035 (0.035) | 3.163 (0.035) | 3.197 (0.035) | 3.179 (0.035) | 3.028 (0.035) | 3.228 (0.035) | 3.208 (0.035) | 3.261 (0.035)

17. Secondary Outcome: Individual PEF Measurements at Each Time Point on Day 29
Description: Adjusted means of the PEF measurements [L/min] at each time point on day 29. Baseline was defined as the mean of the 2 pre-treatment FEV1 values measured on day 1 (-1 hour and -10 minutes) prior to administration of the first dose of study drug.
Time Frame: Baseline and 1 h, 10 min pre-dose and 0 min, 5 min, 30 min, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h post-dose on day 29
Population: FAS
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
L/min
  Timepoint -1:00 hr response | 246.557 (4.061) | 260.901 (4.064) | 263.662 (4.037) | 269.754 (4.110) | 249.356 (4.054) | 263.134 (4.092) | 267.013 (4.064) | 266.913 (4.067)
  Timepoint -0:10 hr response | 245.661 (4.165) | 264.412 (4.180) | 265.177 (4.139) | 271.793 (4.204) | 253.921 (4.157) | 264.808 (4.211) | 268.772 (4.168) | 266.506 (4.183)
  Timepoint 0:00 hr response | 245.758 (3.892) | 262.239 (3.895) | 264.202 (3.870) | 270.565 (3.926) | 251.517 (3.886) | 263.757 (3.921) | 267.623 (3.895) | 266.187 (3.898)
  Timepoint 0:05 hr response | 254.967 (4.259) | 267.969 (4.272) | 273.340 (4.235) | 275.329 (4.307) | 259.301 (4.252) | 271.071 (4.289) | 276.004 (4.262) | 275.727 (4.275)
  Timepoint 0:30 hr response | 257.326 (4.548) | 275.045 (4.563) | 279.309 (4.519) | 286.288 (4.603) | 264.909 (4.539) | 280.836 (4.582) | 287.502 (4.550) | 288.289 (4.566)
  Timepoint 1:00 hr response | 261.890 (4.420) | 279.892 (4.434) | 287.635 (4.393) | 289.866 (4.472) | 263.293 (4.412) | 283.326 (4.452) | 288.427 (4.422) | 288.585 (4.437)
  Timepoint 2:00 hr response | 269.187 (4.606) | 287.181 (4.621) | 295.820 (4.578) | 300.076 (4.661) | 272.318 (4.597) | 291.503 (4.640) | 298.394 (4.609) | 294.627 (4.625)
  Timepoint 3:00 hr response | 269.067 (4.649) | 292.962 (4.665) | 296.736 (4.620) | 303.099 (4.707) | 274.334 (4.641) | 295.008 (4.685) | 296.641 (4.652) | 300.582 (4.669)
  Timepoint 4:00 hr response | 266.451 (4.485) | 286.382 (4.499) | 297.483 (4.460) | 297.415 (4.536) | 274.466 (4.478) | 293.986 (4.517) | 293.617 (4.488) | 302.539 (4.502)
  Timepoint 5:00 hr response | 272.141 (4.500) | 287.917 (4.514) | 293.878 (4.474) | 295.911 (4.550) | 269.220 (4.492) | 293.039 (4.531) | 294.713 (4.502) | 300.335 (4.517)
  Timepoint 6:00 hr response | 268.680 (4.523) | 284.028 (4.537) | 295.843 (4.497) | 295.703 (4.575) | 270.707 (4.515) | 290.283 (4.556) | 293.466 (4.526) | 299.234 (4.541)

18. Secondary Outcome: Weekly Mean Number of Puffs of Rescue Medication Used Per Day
Description: Adjusted means of the weekly mean number of puffs of rescue medication during the whole day : the rescue medication was a salbutamol [albuterol] dose (100 mcg per puff).
Time Frame: Weeks 1 and 4
Population: FAS
Measure: Mean (Standard Error); unit: number of puffs per day
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
number of puffs per day
  Week 1 | 1.511 (0.146) | 1.298 (0.145) | 1.191 (0.147) | 1.446 (0.147) | 1.423 (0.145) | 1.465 (0.147) | 1.172 (0.146) | 1.244 (0.146)
  Week 4 | 1.391 (0.164) | 1.502 (0.163) | 1.299 (0.163) | 1.444 (0.164) | 1.561 (0.162) | 1.344 (0.165) | 1.198 (0.164) | 1.315 (0.163)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.212, 95% CI 2-sided [-0.523 to 0.099], Standard Error of Mean 0.158 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.319, 95% CI 2-sided [-0.634 to -0.004], Standard Error of Mean 0.160 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.065, 95% CI 2-sided [-0.379 to 0.249], Standard Error of Mean 0.160 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.107, 95% CI 2-sided [-0.420 to 0.206], Standard Error of Mean 0.159 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = 0.147, 95% CI 2-sided [-0.168 to 0.462], Standard Error of Mean 0.160 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.255, 95% CI 2-sided [-0.062 to 0.571], Standard Error of Mean 0.161 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.271 to 0.355], Standard Error of Mean 0.160 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.251, 95% CI 2-sided [-0.564 to 0.062], Standard Error of Mean 0.159 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.178, 95% CI 2-sided [-0.492 to 0.135], Standard Error of Mean 0.160 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.293, 95% CI 2-sided [-0.611 to 0.024], Standard Error of Mean 0.162 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.221, 95% CI 2-sided [-0.533 to 0.092], Standard Error of Mean 0.159 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Week 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.073, 95% CI 2-sided [-0.242 to 0.388], Standard Error of Mean 0.160 — Difference calculated as T+O 5/10 minus T+O 2.5/10
Statistical Analysis 13: Comparison: Olo 5 vs T+O 1.25/5; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.110, 95% CI 2-sided [-0.241 to 0.462], Standard Error of Mean 0.179 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 14: Comparison: Olo 5 vs T+O 2.5/5; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.092, 95% CI 2-sided [-0.445 to 0.261], Standard Error of Mean 0.180 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 15: Comparison: Olo 5 vs T+O 5/5; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [-0.301 to 0.406], Standard Error of Mean 0.180 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 16: Comparison: T+O 1.25/5 vs T+O 2.5/5; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.202, 95% CI 2-sided [-0.555 to 0.150], Standard Error of Mean 0.179 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 17: Comparison: T+O 1.25/5 vs T+O 5/5; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.058, 95% CI 2-sided [-0.411 to 0.296], Standard Error of Mean 0.180 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 18: Comparison: T+O 2.5/5 vs T+O 5/5; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.144, 95% CI 2-sided [-0.208 to 0.496], Standard Error of Mean 0.179 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 19: Comparison: Olo 10 vs T+O 1.25/10; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.217, 95% CI 2-sided [-0.568 to 0.135], Standard Error of Mean 0.179 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 20: Comparison: Olo 10 vs T+O 2.5/10; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.363, 95% CI 2-sided [-0.714 to -0.012], Standard Error of Mean 0.179 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 21: Comparison: Olo 10 vs T+O 5/10; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.246, 95% CI 2-sided [-0.598 to 0.106], Standard Error of Mean 0.179 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 22: Comparison: T+O 1.25/10 vs T+O 2.5/10; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.146, 95% CI 2-sided [-0.503 to 0.210], Standard Error of Mean 0.182 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 23: Comparison: T+O 1.25/10 vs T+O 5/10; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.029, 95% CI 2-sided [-0.379 to 0.321], Standard Error of Mean 0.178 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 24: Comparison: T+O 2.5/10 vs T+O 5/10; Week 4; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.117, 95% CI 2-sided [-0.235 to 0.470], Standard Error of Mean 0.180 — Difference calculated as T+O 5/10 minus T+O 2.5/10

19. Secondary Outcome: Physicians Global Evaluation
Description: Adjusted means of the Physicians Global Evaluation of the patient's respiratory condition on days 1 and 29.
  The score was evaluated on a 8-points scale :
  * Poor : 1,2
  * Fair : 3,4
  * Good : 5,6
  * Excellent : 7,8
Time Frame: Days 1 and 29
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
units on a scale
  Day 1 | 4.618 (0.090) | 4.631 (0.090) | 4.484 (0.089) | 4.579 (0.091) | 4.747 (0.090) | 4.464 (0.091) | 4.634 (0.090) | 4.690 (0.090)
  Day 29 | 4.985 (0.093) | 5.146 (0.091) | 5.248 (0.091) | 5.070 (0.094) | 5.109 (0.092) | 5.280 (0.093) | 5.165 (0.092) | 5.227 (0.092)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.014, 95% CI 2-sided [-0.223 to 0.250], Standard Error of Mean 0.121 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.133, 95% CI 2-sided [-0.370 to 0.104], Standard Error of Mean 0.121 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.039, 95% CI 2-sided [-0.278 to 0.199], Standard Error of Mean 0.122 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.147, 95% CI 2-sided [-0.382 to 0.088], Standard Error of Mean 0.120 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.053, 95% CI 2-sided [-0.291 to 0.186], Standard Error of Mean 0.121 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.094, 95% CI 2-sided [-0.144 to 0.332], Standard Error of Mean 0.121 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.282, 95% CI 2-sided [-0.519 to -0.045], Standard Error of Mean 0.121 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.113, 95% CI 2-sided [-0.350 to 0.124], Standard Error of Mean 0.121 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.056, 95% CI 2-sided [-0.293 to 0.180], Standard Error of Mean 0.120 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.169, 95% CI 2-sided [-0.069 to 0.408], Standard Error of Mean 0.121 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.226, 95% CI 2-sided [-0.010 to 0.461], Standard Error of Mean 0.120 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Day 1; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [-0.180 to 0.293], Standard Error of Mean 0.120 — Difference calculated as T+O 5/10 minus T+O 2.5/10
Statistical Analysis 13: Comparison: Olo 5 vs T+O 1.25/5; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.160, 95% CI 2-sided [-0.067 to 0.387], Standard Error of Mean 0.116 — Difference calculated as T+O 1.25/ minus Olo 5
Statistical Analysis 14: Comparison: Olo 5 vs T+O 2.5/5; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.262, 95% CI 2-sided [0.034 to 0.491], Standard Error of Mean 0.116 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 15: Comparison: Olo 5 vs T+O 5/5; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.084, 95% CI 2-sided [-0.148 to 0.316], Standard Error of Mean 0.118 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 16: Comparison: T+O 1.25/5 vs T+O 2.5/5; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [-0.124 to 0.328], Standard Error of Mean 0.115 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 17: Comparison: T+O 1.25/5 vs T+O 5/5; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.076, 95% CI 2-sided [-0.306 to 0.154], Standard Error of Mean 0.117 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 18: Comparison: T+O 2.5/5 vs T+O 5/5; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.178, 95% CI 2-sided [-0.408 to 0.052], Standard Error of Mean 0.117 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 19: Comparison: Olo 10 vs T+O 1.25/10; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.172, 95% CI 2-sided [-0.056 to 0.400], Standard Error of Mean 0.116 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 20: Comparison: Olo 10 vs T+O 2.5/10; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [-0.171 to 0.285], Standard Error of Mean 0.116 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 21: Comparison: Olo 10 vs T+O 5/10; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.118, 95% CI 2-sided [-0.110 to 0.346], Standard Error of Mean 0.116 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 22: Comparison: T+O 1.25/10 vs T+O 2.5/10; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.115, 95% CI 2-sided [-0.345 to 0.115], Standard Error of Mean 0.117 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 23: Comparison: T+O 1.25/10 vs T+O 5/10; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.054, 95% CI 2-sided [-0.281 to 0.173], Standard Error of Mean 0.116 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 24: Comparison: T+O 2.5/10 vs T+O 5/10; Day 29; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.061, 95% CI 2-sided [-0.166 to 0.289], Standard Error of Mean 0.116 — Difference calculated as T+O 5/10 minus T+O 2.5/10

20. Secondary Outcome: Patients Global Rating
Description: Adjusted means of the Global Rating of the patients' health (respiratory condition) on day 29.
  The score was evaluated on a 7-point scale :
  * 1 : very much better
  * 2 : much better
  * 3 : a little better
  * 4 : no change
  * 5 : a little worse
  * 6 : much worse
  * 7 : very much worse
Time Frame: Day 29
Population: FAS
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 107 | 107 | 109 | 104 | 108 | 105 | 107 | 107
units on a scale | 3.357 (0.102) | 3.135 (0.102) | 2.916 (0.102) | 3.208 (0.104) | 3.262 (0.102) | 2.880 (0.103) | 3.130 (0.102) | 2.936 (0.102)
Statistical Analysis 1: Comparison: Olo 5 vs T+O 1.25/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.222, 95% CI 2-sided [-0.481 to 0.037], Standard Error of Mean 0.132 — Difference calculated as T+O 1.25/5 minus Olo 5
Statistical Analysis 2: Comparison: Olo 5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.441, 95% CI 2-sided [-0.700 to -0.182], Standard Error of Mean 0.132 — Difference calculated as T+O 2.5/5 minus Olo 5
Statistical Analysis 3: Comparison: Olo 5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.149, 95% CI 2-sided [-0.409 to 0.111], Standard Error of Mean 0.133 — Difference calculated as T+O 5/5 minus Olo 5
Statistical Analysis 4: Comparison: T+O 1.25/5 vs T+O 2.5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.219, 95% CI 2-sided [-0.478 to 0.040], Standard Error of Mean 0.132 — Difference calculated as T+O 2.5/5 minus T+O 1.25/5
Statistical Analysis 5: Comparison: T+O 1.25/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.073, 95% CI 2-sided [-0.189 to 0.335], Standard Error of Mean 0.133 — Difference calculated as T+O 5/5 minus T+O 1.25/5
Statistical Analysis 6: Comparison: T+O 2.5/5 vs T+O 5/5; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.292, 95% CI 2-sided [0.031 to 0.553], Standard Error of Mean 0.133 — Difference calculated as T+O 5/5 minus T+O 2.5/5
Statistical Analysis 7: Comparison: Olo 10 vs T+O 1.25/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.382, 95% CI 2-sided [-0.641 to -0.123], Standard Error of Mean 0.132 — Difference calculated as T+O 1.25/10 minus Olo 10
Statistical Analysis 8: Comparison: Olo 10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.132, 95% CI 2-sided [-0.390 to 0.127], Standard Error of Mean 0.132 — Difference calculated as T+O 2.5/10 minus Olo 10
Statistical Analysis 9: Comparison: Olo 10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.326, 95% CI 2-sided [-0.585 to -0.067], Standard Error of Mean 0.132 — Difference calculated as T+O 5/10 minus Olo 10
Statistical Analysis 10: Comparison: T+O 1.25/10 vs T+O 2.5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.250, 95% CI 2-sided [-0.010 to 0.511], Standard Error of Mean 0.133 — Difference calculated as T+O 2.5/10 minus T+O 1.25/10
Statistical Analysis 11: Comparison: T+O 1.25/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.056, 95% CI 2-sided [-0.202 to 0.314], Standard Error of Mean 0.132 — Difference calculated as T+O 5/10 minus T+O 1.25/10
Statistical Analysis 12: Comparison: T+O 2.5/10 vs T+O 5/10; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = -0.194, 95% CI 2-sided [-0.453 to 0.065], Standard Error of Mean 0.132 — Difference calculated as T+O 5/10 minus T+O 2.5/10

21. Secondary Outcome: Pulse Rate Recorded in Conjunction With Spirometry
Description: Pulse rate recorded in conjunction with spirometry change from baseline at 30 minutes post-dose on day 29 in beats per minute (bpm).
Time Frame: Baseline and 30 min post-dose on day 29
Population: TS which comprised all patients who were dispensed study medication, were documented to have taken at least 1 dose of investigational treatment and had available data for pulse rate at baseline and day 29.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 105 | 105 | 111 | 106 | 108 | 106 | 108 | 107
bpm | -2.4 (10.4) | -2.8 (10.3) | -3.1 (10.3) | -1.8 (9.5) | -2.1 (8.5) | -3.6 (9.6) | -2.4 (10.5) | -1.0 (10.2)

22. Secondary Outcome: Systolic and Diastolic Blood Pressure Recorded in Conjunction With Spirometry
Description: Systolic and diastolic blood pressure recorded in conjunction with spirometry change from baseline on day 29 in millimetres of mercury (mmHg).
Time Frame: Baseline and 30 min post-dose on day 29
Population: TS which comprised all patients who were dispensed study medication, were documented to have taken at least 1 dose of investigational treatment and had available data for systolic and diastolic blood pressure at baseline and day 29.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Number analyzed (Participants) | 105 | 105 | 111 | 106 | 108 | 106 | 108 | 107
mmHg
  Systolic blood pressure | -7.2 (15.0) | -6.0 (12.8) | -5.6 (15.0) | -4.8 (13.9) | -3.4 (14.7) | -5.5 (15.2) | -3.8 (14.2) | -2.2 (13.0)
  Diastolic blood pressure | -3.8 (9.1) | -2.8 (8.6) | -2.5 (9.8) | -3.0 (9.8) | -3.0 (8.6) | -3.0 (9.1) | -2.5 (9.7) | -0.4 (9.2)

ADVERSE EVENTS:
Time Frame: From first drug administration until 21 days after the last administration, up to 75 days
Arm/Group | Olo 5 | T+O 1.25/5 | T+O 2.5/5 | T+O 5/5 | Olo 10 | T+O 1.25/10 | T+O 2.5/10 | T+O 5/10
Serious Adverse Events (participants affected / at risk) | 4/108 | 1/109 | 3/113 | 1/109 | 2/109 | 1/110 | 5/110 | 0/111
Other Adverse Events (participants affected / at risk) | 15/108 | 15/109 | 11/113 | 11/109 | 12/109 | 13/110 | 7/110 | 6/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olo 5 (N=108) | T+O 1.25/5 (N=109) | T+O 2.5/5 (N=113) | T+O 5/5 (N=109) | Olo 10 (N=109) | T+O 1.25/10 (N=110) | T+O 2.5/10 (N=110) | T+O 5/10 (N=111)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olo 5 (N=108) | T+O 1.25/5 (N=109) | T+O 2.5/5 (N=113) | T+O 5/5 (N=109) | Olo 10 (N=109) | T+O 1.25/10 (N=110) | T+O 2.5/10 (N=110) | T+O 5/10 (N=111)
Nasopharyngitis (Infections and infestations) | 11 | 12 | 8 | 3 | 7 | 8 | 4 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 3 | 8 | 6 | 7 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.